CLINICAL TRIAL: NCT06790927
Title: A Cluster Randomized Controlled Trial on a Standardized Antihypertensive Treatment Protocol
Brief Title: Standardized Antihypertensive Treatment Protocol
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Vital Strategies (Other)
Responsible Party: Principal Investigator, Ji-Guang Wang, Prof, Shanghai Institute of Hypertension
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Standardized Protocol
Record Dates: First submitted 2025-01-14; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Eligible patients will be divided into two groups. In the usual treatment group, the doctor prescribes medication for patients, and advise the patient to take the medication on time and follow-up every 3 months. The standard treatment group was followed up monthly, Amlodipine 5 mg is preferred for selected patients, and amlodipine 5 mg + irbesartan 150mg is used for those who do not meet blood pressure targets after 4 weeks treatment, amlodipine 10mg + irbesartan 300mg is used for those who do not meet blood pressure targets after one month, for those whose blood pressure is still not up to standard after 4 weeks will be treated with amlodipine 10mg + irbesartan 300mg + hydrochlorothiazide 12.5mg
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- usual treatment group (Active Comparator)
  Interventions: Drug: Usual Care
- standard treatment group (Experimental)
  Interventions: Drug: Standard Medical Therapy

INTERVENTIONS:
Drug: Usual Care — The doctor prescribes medication for patients and follow-up every 3 months
  Arms: usual treatment group
Drug: Standard Medical Therapy — The standard treatment group was followed up monthly, Amlodipine 5 mg is preferred for selected patients, and amlodipine 5 mg + irbesartan 150mg is used for those who do not meet blood pressure targets after 4 weeks treatment, amlodipine 10mg + irbesartan 300mg is used for those who do not meet blood pressure targets after one month, for those whose blood pressure is still not up to standard after 4 weeks will be treated with amlodipine 10mg + irbesartan 300mg + hydrochlorothiazide 12.5mg.
  Arms: standard treatment group

SUMMARY:
Study name: A cluster randomized controlled trial on a standardized antihypertensive treatment protocol.

Objective: To evaluate a simple treatment protocol for China in a real clinic setting.

Study design: In this study, newly identified uncontrolled hypertension or monotherapy for patients with substandard blood pressure are sequentially enrolled and monitored for blood pressure in the office and at home. Randomization was carried out on a machine numeric table, one center with a small value assigned to the usual care group and one with a larger number was assigned to the standard treatment group.

Study population: Men and Women aged 18-80 years (n=400) meeting the inclusion/exclusion criteria.

Randomization and treatment: Randomization was carried out on a machine numeric table, one center with a small value assigned to the usual care group and one with a larger number was assigned to the standard treatment group. In the usual treatment group, the doctor prescribes medication for patients, and advise the patient to take the medication on time and follow-up every 3 months. The standard treatment group was followed up monthly, Amlodipine 5 mg is preferred for selected patients, and amlodipine 5 mg + irbesartan 150mg is used for those who do not meet blood pressure targets after 4 weeks of treatment, aftre one month amlodipine 10mg + irbesartan 300mg is used for those who do not meet blood pressure targets, for those whose blood pressure is still not up to standard after 4 weeks will be treated with amlodipine 10mg + irbesartan 300mg + hydrochlorothiazide 12.5mg.

Follow up: 6 months. Sample size: a total of 400 patients should be enrolled in the combination. Timeline: After obtaining the approval of Ethics Committee of Ruijin Hospital in November 2024, Patients enrollment will be performed between Feburary 2025 to Feburary 2026.

DETAILED DESCRIPTION:
Study name: A cluster randomized controlled trial on a standardized antihypertensive treatment protocol.

Objective: To evaluate a simple treatment protocol for China in a real clinic setting.

Study design: In this study, newly identified uncontrolled hypertension or monotherapy for patients with substandard blood pressure are sequentially enrolled and monitored for blood pressure in the office and at home. Randomization was carried out on a machine numeric table, one center with a small value assigned to the usual care group and one with a larger number was assigned to the standard treatment group.

Study population: Men and Women aged 18-80 years (n=400) meeting the inclusion/exclusion criteria. Inclusion Criteria: (1) Age 18-80 years; (2) Newly identified or monotherapy patients with uncontrolled clinical blood pressure; (3) Systolic blood pressure≥140 mmHg and/or diastolic blood pressure≥90 mmHg; (4) Agree to participate in the trial and sign the informed consent form. Exclusion criteria: (1) The arm circumference is too large or too small (<17cm or >42cm) ; (2) suspected or definite secondary hypertension; (3) Combined with eGFR < 30 ml/min/1.73m2 or end-stage renal disease; (4) Cardiovascular and cerebrovascular events have occurred in the past 3 months, such as myocardial infarction, stroke, acute heart failure, causes Unstable angina pectoris, hospitalization or revascularization of coronary artery disease or bypass graft surgery; (5) Combined with liver damage: aspartate aminotransferase [AST] or alanine aminotransferase [ALT] or total bilirubin at 2 times or more of the upper limit of normal; (6) Concomitant physical diseases with survival expectations of less than 3 years, or tumors diagnosed in the past 2 years and requiring treatment; (7) The investigator assessed that participation in the study was unfavorable to the subject.

Randomization and treatment: Randomization was carried out on a machine numeric table, one center with a small value assigned to the usual care group and one with a larger number was assigned to the standard treatment group. In the usual treatment group, the doctor prescribes medication for patients, and advise the patient to take the medication on time and follow-up every 3 months. The standard treatment group was followed up monthly, Amlodipine 5 mg is preferred for selected patients, and amlodipine 5 mg + irbesartan 150mg is used for those who do not meet blood pressure targets after 4 weeks of treatment, aftre one month amlodipine 10mg + irbesartan 300mg is used for those who do not meet blood pressure targets, for those whose blood pressure is still not up to standard after 4 weeks will be treated with amlodipine 10mg + irbesartan 300mg + hydrochlorothiazide 12.5mg.

Follow up: 6 months. Sample size: At least 200 eligible patients should be enrolled in each group, a total of 400 patients should be enrolled in the combination.

Timeline: After obtaining the approval of Ethics Committee of Ruijin Hospital in November 2024, Patients enrollment will be performed between Feburary 2025 to Feburary 2026. Database construction and statistical analysis will be conducted at the same time, appropriate domestic and international conferences will be selected to publish the research results. The main results will be published in international professional medical journals.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years;
2. Newly identified or monotherapy patients with uncontrolled clinical blood pressure;
3. Systolic blood pressure≥140 mmHg and/or diastolic blood pressure≥90 mmHg;
4. Agree to participate in the trial and sign the informed consent form.

Exclusion criteria:

1. The arm circumference is too large or too small (<17cm or >42cm) ;
2. suspected or definite secondary hypertension;
3. Combined with eGFR < 30 ml/min/1.73m2 or end-stage renal disease;
4. Cardiovascular and cerebrovascular events have occurred in the past 3 months, such as myocardial infarction, stroke, acute heart failure, causes Unstable angina pectoris, hospitalization or revascularization of coronary artery disease or bypass graft surgery;
5. Combined with liver damage: aspartate aminotransferase [AST] or alanine aminotransferase [ALT] or total bilirubin at 2 times or more of the upper limit of normal;
6. Concomitant physical diseases with survival expectations of less than 3 years, or tumors diagnosed in the past 2 years and requiring treatment;
7. The investigator assessed that participation in the study was unfavorable to the subject.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-02-24 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Control rate of clinical blood pressure | 6 months

SECONDARY OUTCOMES:
Control rate of home blood pressure | 6 months
The rate at which doctor prescribe according to standard treatment protocol | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Institute of Hypertension, Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, China, China